CLINICAL TRIAL: NCT06429293
Title: Impact of Cognitive Behavioral Therapy on Neural, Inflammatory, & Autonomic Markers in a Sample With PTSD and Cardiovascular Risk: Protocol for a Pilot Randomized Controlled Trial
Brief Title: Impact of Cognitive Behavioral Therapy on PTSD-CVD Link
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Michael T. Osborne, Clinician Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023P001621
Record Dates: First submitted 2024-05-08; First posted 2024-05-24 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Cardiovascular disease; Inflammation; Autonomic function; Stress-related neural activity
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Intervention Model Description: Participants are randomized to 12 weeks of cognitive processing therapy or waitlist control.
Who Masked: Outcomes Assessor
Masking Description: Individuals who interpret images and data will be blinded to assigned intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive processing therapy (Experimental): 12 week treatment period of cognitive processing therapy followed by a post-treatment visit.
  Interventions: Behavioral: Cognitive processing therapy
- Control waitlist (No Intervention): Participants randomized to waitlist are offered CPT upon completion of the post-treatment visit.

INTERVENTIONS:
Behavioral: Cognitive processing therapy — The active intervention is Cognitive Processing Therapy (CPT) is a gold-standard cognitive behavioral therapy for PTSD. The CPT intervention consists of 12 60-minute sessions teaching skills to challenge trauma-relevant cognitions that are distorted or unhelpful. Trauma-relevant cognitions fall into five themes that are highlighted during treatment: safety, trust, power/control, esteem, and intimacy. The empirical base for CPT is strong with numerous studies demonstrating that it results in significant reduction of PTSD symptoms regardless of trauma type and that it is 89% more effective than control treatment. CPT has been successfully implemented in virtual formats with comparable efficacy levels to that of in-person CPT. CPT sessions for this study will be conducted virtually by a CPT-trained clinician
  Arms: Cognitive processing therapy

SUMMARY:
This is a pilot randomized controlled trial to assess the impact of a first-line treatment for posttraumatic stress disorder (PTSD) (Cognitive Processing Therapy; CPT) versus waitlist control on mechanisms of cardiovascular disease (CVD) risk. Further, this study will test the hypothesis that CPT reduces CVD risk through its effects on inflammation and autonomic function and that these changes are driven by changes in stress-related neural activity (SNA)

DETAILED DESCRIPTION:
This study is a randomized controlled trial of CPT compared to waitlist control that is testing the effects of CPT on mechanisms of the PTSD-CVD link. Enrollment began in 2023 and is projected to continue through 2026. Participants include individuals with PTSD and CVD risk recruited from the Boston area (N = 30). Treatment assignment is randomized and stratified by sex. Participants are randomized to CPT (n = 15) or waitlist control (n = 15). Potentially eligible participants complete a screening visit to confirm inclusion/exclusion criteria. Upon confirmation of eligibility, participants are scheduled for a baseline session, where they complete surveys, brain and peripheral imaging, and resting measures of autonomic function. Following the baseline visit, participants are randomized into CPT or the waitlist control group. Those randomized to CPT complete sessions via telehealth. Following a 12-week treatment period, participants attend the post-treatment visit, consisting of the same assessments administered at baseline. Participants randomized to waitlist are offered CPT upon completion of the post-treatment visit.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years (upper limit chosen to optimize changes in brain activation that diminish with age);
* criterion A trauma exposure and PTSD symptoms (clinically significant symptoms in at least two symptom clusters);
* subclinical atherosclerotic CVD (e.g., coronary, cerebrovascular, or peripheral arterial plaque or calcifications on imaging), clinical atherosclerotic CVD (e.g., myocardial infarction or revascularization), or increased risk for atherosclerotic CVD (i.e., >2 of hypertension, diabetes mellitus, hyperlipidemia, and active smoking) ability to understand and sign informed consent
* fluent English speaker.

Exclusion Criteria:

* history of stroke, brain surgery, seizure
* use of certain CVD medications (e.g., beta-blockers, high-intensity statins [e.g., rosuvastatin 20/40 mg and atorvastatin 40/80 mg], PCSK-9 inhibitors);
* psychiatric or cardiovascular medication change within 4 weeks (i.e., stable regimen is allowed);
* currently in PTSD therapy;
* neurological or systemic inflammatory disease/current anti-inflammatory therapy;
* moderate/severe alcohol/substance use disorder;
* current mania/psychosis;
* weight >300 lbs., claustrophobia, pregnancy, metal implants that are incompatible with magnetic resonance imaging (MRI), or uncontrolled hyperglycemia (for imaging);
* significant radiation exposure (>2 nuclear tests, computed tomography images, or fluoroscopic procedures) for research purposes during the preceding 12-months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Arterial inflammation | Baseline and 12-weeks
  Measured via FDG-PET imaging
Heart rate variability | Baseline and 12-weeks
  Calculated from the average resting HRV collected at baseline and post-treatment visits

SECONDARY OUTCOMES:
Leukopoiesis | Baseline and 12-weeks
  Measured as bone marrow activity via FDG-PET imaging
Heart rate | Baseline and 12-weeks
  Heart rate in beats per minute
Blood pressure | Baseline and 12-weeks
  Systolic and diastolic pressure
MRI based arterial plaque components (such as necrotic tissue, loose connective tissue, and hemorrhage) | Baseline and 12-weeks
  MRI measurements of atherosclerotic plaque components including necrotic tissue, loose connective tissue, and hemorrhage using black-blood imaging techniques
MRI based arterial wall thickness | Baseline and 12-weeks
  Measurements of wall thickness as an assessment of atherosclerotic plaque
MRI based brain structure assessments of volume and density | Baseline and 12-weeks
  Structural assessment of brain centers to assess volume and density of neural centers involved in the stress response
MRI based brain connectivity (by measuring changes in blood flow across networks of neural centers at rest and with an emotional task) | Baseline and 12-weeks
  Connectivity assessment using mapping on functional MRI at baseline and in response to emotional faces of neural centers involved in the stress response to determine the interplay between neural centers before and after therapy by measuring alterations in blood oxygen content under various conditions in different parts of the brain
MRI based brain activation (via measuring blood flow in important neural centers at rest and with an emotional task using functional MRI) | Baseline and 12-weeks
  Activation assessment using functional MRI at both rest and in response to emotional faces of neural centers involved in the stress response before and after therapy by measuring blood flow under various conditions to different parts of the brain
Axonal integrity of resting neural connections between brain centers using MRI | Baseline and 12-weeks
  Measurement of axonal integrity using diffusion tensor imaging on MRI to determine the strength connections between important brain centers and neural networks related to stress perception in PTSD before and after therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data from primary endpoints and analyses will be made available on a public website following study completion.
Time Frame: Within 6 months of study completion
Access Criteria: To be determined based on website used

REFERENCES:
- [Background] Edmondson D, Cohen BE. Posttraumatic stress disorder and cardiovascular disease. Prog Cardiovasc Dis. 2013 May-Jun;55(6):548-56. doi: 10.1016/j.pcad.2013.03.004. Epub 2013 Apr 6. PMID 23621964
- [Background] Edmondson D, von Kanel R. Post-traumatic stress disorder and cardiovascular disease. Lancet Psychiatry. 2017 Apr;4(4):320-329. doi: 10.1016/S2215-0366(16)30377-7. Epub 2017 Jan 19. PMID 28109646
- [Background] Kessler RC, Sonnega A, Bromet E, Hughes M, Nelson CB. Posttraumatic stress disorder in the National Comorbidity Survey. Arch Gen Psychiatry. 1995 Dec;52(12):1048-60. doi: 10.1001/archpsyc.1995.03950240066012. PMID 7492257
- [Background] Goldstein RB, Smith SM, Chou SP, Saha TD, Jung J, Zhang H, Pickering RP, Ruan WJ, Huang B, Grant BF. The epidemiology of DSM-5 posttraumatic stress disorder in the United States: results from the National Epidemiologic Survey on Alcohol and Related Conditions-III. Soc Psychiatry Psychiatr Epidemiol. 2016 Aug;51(8):1137-48. doi: 10.1007/s00127-016-1208-5. Epub 2016 Apr 22. PMID 27106853
- [Background] Ehlers A, Suendermann O, Boellinghaus I, Vossbeck-Elsebusch A, Gamer M, Briddon E, Martin MW, Glucksman E. Heart rate responses to standardized trauma-related pictures in acute posttraumatic stress disorder. Int J Psychophysiol. 2010 Oct;78(1):27-34. doi: 10.1016/j.ijpsycho.2010.04.009. Epub 2010 May 5. PMID 20450940
- [Background] Jovanovic T, Norrholm SD, Sakoman AJ, Esterajher S, Kozaric-Kovacic D. Altered resting psychophysiology and startle response in Croatian combat veterans with PTSD. Int J Psychophysiol. 2009 Mar;71(3):264-8. doi: 10.1016/j.ijpsycho.2008.10.007. Epub 2008 Nov 5. PMID 19013485
- [Background] Buckley TC, Kaloupek DG. A meta-analytic examination of basal cardiovascular activity in posttraumatic stress disorder. Psychosom Med. 2001 Jul-Aug;63(4):585-94. doi: 10.1097/00006842-200107000-00011. PMID 11485112
- [Background] Pan X, Kaminga AC, Wen SW, Liu A. Catecholamines in Post-traumatic Stress Disorder: A Systematic Review and Meta-Analysis. Front Mol Neurosci. 2018 Dec 4;11:450. doi: 10.3389/fnmol.2018.00450. eCollection 2018. PMID 30564100
- [Background] Brudey C, Park J, Wiaderkiewicz J, Kobayashi I, Mellman TA, Marvar PJ. Autonomic and inflammatory consequences of posttraumatic stress disorder and the link to cardiovascular disease. Am J Physiol Regul Integr Comp Physiol. 2015 Aug 15;309(4):R315-21. doi: 10.1152/ajpregu.00343.2014. Epub 2015 Jun 10. PMID 26062635
- [Background] Kim TD, Lee S, Yoon S. Inflammation in Post-Traumatic Stress Disorder (PTSD): A Review of Potential Correlates of PTSD with a Neurological Perspective. Antioxidants (Basel). 2020 Jan 26;9(2):107. doi: 10.3390/antiox9020107. PMID 31991875
- [Background] Schneider M, Schwerdtfeger A. Autonomic dysfunction in posttraumatic stress disorder indexed by heart rate variability: a meta-analysis. Psychol Med. 2020 Sep;50(12):1937-1948. doi: 10.1017/S003329172000207X. Epub 2020 Aug 28. PMID 32854795
- [Background] Ge F, Yuan M, Li Y, Zhang W. Posttraumatic Stress Disorder and Alterations in Resting Heart Rate Variability: A Systematic Review and Meta-Analysis. Psychiatry Investig. 2020 Jan;17(1):9-20. doi: 10.30773/pi.2019.0112. Epub 2020 Jan 25. PMID 31995968
- [Background] Moon E, Lee SH, Kim DH, Hwang B. Comparative Study of Heart Rate Variability in Patients with Schizophrenia, Bipolar Disorder, Post-traumatic Stress Disorder, or Major Depressive Disorder. Clin Psychopharmacol Neurosci. 2013 Dec;11(3):137-43. doi: 10.9758/cpn.2013.11.3.137. Epub 2013 Dec 24. PMID 24465250
- [Background] Seligowski AV, Steuber ER, Hinrichs R, Reda MH, Wiltshire CN, Wanna CP, Winters SJ, Phillips KA, House SL, Beaudoin FL, An X, Stevens JS, Zeng D, Neylan TC, Clifford GD, Linnstaedt SD, Germine LT, Bollen KA, Guffanti G, Rauch SL, Haran JP, Storrow AB, Lewandowski C, Musey PI Jr, Hendry PL, Sheikh S, Jones CW, Punches BE, Kurz MC, Murty VP, McGrath ME, Hudak LA, Pascual JL, Seamon MJ, Datner EM, Chang AM, Pearson C, Peak DA, Merchant RC, Domeier RM, Rathlev NK, O'Neil BJ, Sanchez LD, Bruce SE, Miller MW, Pietrzak RH, Joormann J, Barch DM, Pizzagalli DA, Sheridan JF, Luna B, Harte SE, Elliott JM, Koenen KC, Kessler RC, McLean SA, Ressler KJ, Jovanovic T. A prospective examination of sex differences in posttraumatic autonomic functioning. Neurobiol Stress. 2021 Aug 21;15:100384. doi: 10.1016/j.ynstr.2021.100384. eCollection 2021 Nov. PMID 34485632
- [Background] Seligowski AV, Grewal SS, Abohashem S, Zureigat H, Qamar I, Aldosoky W, Gharios C, Hanlon E, Alani O, Bollepalli SC, Armoundas A, Fayad ZA, Shin LM, Osborne MT, Tawakol A. PTSD increases risk for major adverse cardiovascular events through neural and cardio-inflammatory pathways. Brain Behav Immun. 2024 Mar;117:149-154. doi: 10.1016/j.bbi.2024.01.006. Epub 2024 Jan 11. PMID 38218349
- [Background] O'Donovan A, Neylan TC, Metzler T, Cohen BE. Lifetime exposure to traumatic psychological stress is associated with elevated inflammation in the Heart and Soul Study. Brain Behav Immun. 2012 May;26(4):642-9. doi: 10.1016/j.bbi.2012.02.003. Epub 2012 Feb 15. PMID 22366689
- [Background] Tawakol A, Ishai A, Takx RA, Figueroa AL, Ali A, Kaiser Y, Truong QA, Solomon CJ, Calcagno C, Mani V, Tang CY, Mulder WJ, Murrough JW, Hoffmann U, Nahrendorf M, Shin LM, Fayad ZA, Pitman RK. Relation between resting amygdalar activity and cardiovascular events: a longitudinal and cohort study. Lancet. 2017 Feb 25;389(10071):834-845. doi: 10.1016/S0140-6736(16)31714-7. Epub 2017 Jan 12. PMID 28088338
- [Background] Lima BB, Hammadah M, Wilmot K, Pearce BD, Shah A, Levantsevych O, Kaseer B, Obideen M, Gafeer MM, Kim JH, Sullivan S, Lewis TT, Weng L, Elon L, Li L, Bremner JD, Raggi P, Quyyumi A, Vaccarino V. Posttraumatic stress disorder is associated with enhanced interleukin-6 response to mental stress in subjects with a recent myocardial infarction. Brain Behav Immun. 2019 Jan;75:26-33. doi: 10.1016/j.bbi.2018.08.015. Epub 2018 Aug 30. PMID 30172946
- [Background] Myers B. Corticolimbic regulation of cardiovascular responses to stress. Physiol Behav. 2017 Apr 1;172:49-59. doi: 10.1016/j.physbeh.2016.10.015. Epub 2016 Oct 25. PMID 27793557
- [Background] Shin LM, Orr SP, Carson MA, Rauch SL, Macklin ML, Lasko NB, Peters PM, Metzger LJ, Dougherty DD, Cannistraro PA, Alpert NM, Fischman AJ, Pitman RK. Regional cerebral blood flow in the amygdala and medial prefrontal cortex during traumatic imagery in male and female Vietnam veterans with PTSD. Arch Gen Psychiatry. 2004 Feb;61(2):168-76. doi: 10.1001/archpsyc.61.2.168. PMID 14757593
- [Background] Shin LM, Wright CI, Cannistraro PA, Wedig MM, McMullin K, Martis B, Macklin ML, Lasko NB, Cavanagh SR, Krangel TS, Orr SP, Pitman RK, Whalen PJ, Rauch SL. A functional magnetic resonance imaging study of amygdala and medial prefrontal cortex responses to overtly presented fearful faces in posttraumatic stress disorder. Arch Gen Psychiatry. 2005 Mar;62(3):273-81. doi: 10.1001/archpsyc.62.3.273. PMID 15753240
- [Background] Williams LM, Kemp AH, Felmingham K, Barton M, Olivieri G, Peduto A, Gordon E, Bryant RA. Trauma modulates amygdala and medial prefrontal responses to consciously attended fear. Neuroimage. 2006 Jan 15;29(2):347-57. doi: 10.1016/j.neuroimage.2005.03.047. Epub 2005 Oct 10. PMID 16216534
- [Background] Stevens JS, Jovanovic T, Fani N, Ely TD, Glover EM, Bradley B, Ressler KJ. Disrupted amygdala-prefrontal functional connectivity in civilian women with posttraumatic stress disorder. J Psychiatr Res. 2013 Oct;47(10):1469-78. doi: 10.1016/j.jpsychires.2013.05.031. Epub 2013 Jul 1. PMID 23827769
- [Background] Osborne MT, Abohashem S, Zureigat H, Abbasi TA, Tawakol A. Multimodality molecular imaging: Gaining insights into the mechanisms linking chronic stress to cardiovascular disease. J Nucl Cardiol. 2021 Jun;28(3):955-966. doi: 10.1007/s12350-020-02424-6. Epub 2020 Nov 17. PMID 33205328
- [Background] Manthey A, Sierk A, Brakemeier EL, Walter H, Daniels JK. Does trauma-focused psychotherapy change the brain? A systematic review of neural correlates of therapeutic gains in PTSD. Eur J Psychotraumatol. 2021 Aug 6;12(1):1929025. doi: 10.1080/20008198.2021.1929025. eCollection 2021. PMID 34394855
- [Background] Aupperle RL, Allard CB, Simmons AN, Flagan T, Thorp SR, Norman SB, Paulus MP, Stein MB. Neural responses during emotional processing before and after cognitive trauma therapy for battered women. Psychiatry Res. 2013 Oct 30;214(1):48-55. doi: 10.1016/j.pscychresns.2013.05.001. Epub 2013 Aug 2. PMID 23916537
- [Background] Santarnecchi E, Bossini L, Vatti G, Fagiolini A, La Porta P, Di Lorenzo G, Siracusano A, Rossi S, Rossi A. Psychological and Brain Connectivity Changes Following Trauma-Focused CBT and EMDR Treatment in Single-Episode PTSD Patients. Front Psychol. 2019 Feb 25;10:129. doi: 10.3389/fpsyg.2019.00129. eCollection 2019. PMID 30858808
- [Background] Helpman L, Marin MF, Papini S, Zhu X, Sullivan GM, Schneier F, Neria M, Shvil E, Malaga Aragon MJ, Markowitz JC, Lindquist MA, Wager T, Milad M, Neria Y. Neural changes in extinction recall following prolonged exposure treatment for PTSD: A longitudinal fMRI study. Neuroimage Clin. 2016 Oct 10;12:715-723. doi: 10.1016/j.nicl.2016.10.007. eCollection 2016. PMID 27761402
- [Background] Zhu X, Suarez-Jimenez B, Lazarov A, Helpman L, Papini S, Lowell A, Durosky A, Lindquist MA, Markowitz JC, Schneier F, Wager TD, Neria Y. Exposure-based therapy changes amygdala and hippocampus resting-state functional connectivity in patients with posttraumatic stress disorder. Depress Anxiety. 2018 Oct;35(10):974-984. doi: 10.1002/da.22816. Epub 2018 Sep 10. PMID 30260530
- [Background] Abdallah CG, Averill CL, Ramage AE, Averill LA, Alkin E, Nemati S, Krystal JH, Roache JD, Resick P, Young-McCaughan S, Peterson AL, Fox P; STRONG STAR Consortium. Reduced Salience and Enhanced Central Executive Connectivity Following PTSD Treatment. Chronic Stress (Thousand Oaks). 2019 Jan-Feb;3:2470547019838971. doi: 10.1177/2470547019838971. Epub 2019 Apr 15. PMID 31008419
- [Background] Watkins LL, LoSavio ST, Calhoun P, Resick PA, Sherwood A, Coffman CJ, Kirby AC, Beaver TA, Dennis MF, Beckham JC. Effect of cognitive processing therapy on markers of cardiovascular risk in posttraumatic stress disorder patients: A randomized clinical trial. J Psychosom Res. 2023 Jul;170:111351. doi: 10.1016/j.jpsychores.2023.111351. Epub 2023 May 2. PMID 37178469
- [Background] Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess. 2018 Mar;30(3):383-395. doi: 10.1037/pas0000486. Epub 2017 May 11. PMID 28493729
- [Background] Radfar A, Abohashem S, Osborne MT, Wang Y, Dar T, Hassan MZO, Ghoneem A, Naddaf N, Patrich T, Abbasi T, Zureigat H, Jaffer J, Ghazi P, Scott JA, Shin LM, Pitman RK, Neilan TG, Wood MJ, Tawakol A. Stress-associated neurobiological activity associates with the risk for and timing of subsequent Takotsubo syndrome. Eur Heart J. 2021 May 14;42(19):1898-1908. doi: 10.1093/eurheartj/ehab029. PMID 33768230
- [Background] Emami H, Singh P, MacNabb M, Vucic E, Lavender Z, Rudd JH, Fayad ZA, Lehrer-Graiwer J, Korsgren M, Figueroa AL, Fredrickson J, Rubin B, Hoffmann U, Truong QA, Min JK, Baruch A, Nasir K, Nahrendorf M, Tawakol A. Splenic metabolic activity predicts risk of future cardiovascular events: demonstration of a cardiosplenic axis in humans. JACC Cardiovasc Imaging. 2015 Feb;8(2):121-30. doi: 10.1016/j.jcmg.2014.10.009. Epub 2015 Jan 7. PMID 25577441
- [Background] Hariri AR, Bookheimer SY, Mazziotta JC. Modulating emotional responses: effects of a neocortical network on the limbic system. Neuroreport. 2000 Jan 17;11(1):43-8. doi: 10.1097/00001756-200001170-00009. PMID 10683827
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Asmundson GJG, Thorisdottir AS, Roden-Foreman JW, Baird SO, Witcraft SM, Stein AT, Smits JAJ, Powers MB. A meta-analytic review of cognitive processing therapy for adults with posttraumatic stress disorder. Cogn Behav Ther. 2019 Jan;48(1):1-14. doi: 10.1080/16506073.2018.1522371. Epub 2018 Oct 18. PMID 30332919
- [Background] Kline AC, Cooper AA, Rytwinksi NK, Feeny NC. Long-term efficacy of psychotherapy for posttraumatic stress disorder: A meta-analysis of randomized controlled trials. Clin Psychol Rev. 2018 Feb;59:30-40. doi: 10.1016/j.cpr.2017.10.009. Epub 2017 Nov 21. PMID 29169664
- [Background] Watts BV, Schnurr PP, Mayo L, Young-Xu Y, Weeks WB, Friedman MJ. Meta-analysis of the efficacy of treatments for posttraumatic stress disorder. J Clin Psychiatry. 2013 Jun;74(6):e541-50. doi: 10.4088/JCP.12r08225. PMID 23842024
- [Background] Held P, Kovacevic M, Petrey K, Meade EA, Pridgen S, Montes M, Werner B, Miller ML, Smith DL, Kaysen D, Karnik NS. Treating posttraumatic stress disorder at home in a single week using 1-week virtual massed cognitive processing therapy. J Trauma Stress. 2022 Aug;35(4):1215-1225. doi: 10.1002/jts.22831. Epub 2022 Mar 25. PMID 35338534
- [Background] Held P, Coleman JA, Petrey K, Klassen BJ, Pridgen S, Bravo K, Smith DL, Van Horn R. A case series examining PTSD and depression symptom reductions over the course of a 2-week virtual intensive PTSD treatment program for veterans. Psychol Trauma. 2022 May;14(4):615-623. doi: 10.1037/tra0001106. Epub 2021 Aug 26. PMID 34435816
- [Background] Tawakol A, Fayad ZA, Mogg R, Alon A, Klimas MT, Dansky H, Subramanian SS, Abdelbaky A, Rudd JH, Farkouh ME, Nunes IO, Beals CR, Shankar SS. Intensification of statin therapy results in a rapid reduction in atherosclerotic inflammation: results of a multicenter fluorodeoxyglucose-positron emission tomography/computed tomography feasibility study. J Am Coll Cardiol. 2013 Sep 3;62(10):909-17. doi: 10.1016/j.jacc.2013.04.066. Epub 2013 May 30. PMID 23727083
- [Background] Bourassa KJ, Hendrickson RC, Reger GM, Norr AM. Posttraumatic Stress Disorder Treatment Effects on Cardiovascular Physiology: A Systematic Review and Agenda for Future Research. J Trauma Stress. 2021 Apr;34(2):384-393. doi: 10.1002/jts.22637. Epub 2020 Dec 5. PMID 33277952
- [Background] Gan WQ, Buxton JA, Scheuermeyer FX, Palis H, Zhao B, Desai R, Janjua NZ, Slaunwhite AK. Risk of cardiovascular diseases in relation to substance use disorders. Drug Alcohol Depend. 2021 Dec 1;229(Pt A):109132. doi: 10.1016/j.drugalcdep.2021.109132. Epub 2021 Oct 27. PMID 34768052
- [Background] Byers AL, Covinsky KE, Neylan TC, Yaffe K. Chronicity of posttraumatic stress disorder and risk of disability in older persons. JAMA Psychiatry. 2014 May;71(5):540-6. doi: 10.1001/jamapsychiatry.2014.5. PMID 24647756
- [Background] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Derived] Ellis R, Sinnott S, Karam K, Assefa A, Osborne M, Seligowski A. Impact of cognitive behavioural therapy on neural, inflammatory, & autonomic markers in a sample with PTSD and cardiovascular risk: protocol for a pilot randomised controlled trial. Eur J Psychotraumatol. 2024;15(1):2378618. doi: 10.1080/20008066.2024.2378618. Epub 2024 Jul 24. PMID 39045795
- See also: About Multiple Cause of Death — https://wonder.cdc.gov/mcd-icd10.html
- See also: The Life Events Checklist for DSM-5 (LEC-5) — https://www.ptsd.va.gov/professional/assessment/te-measures/life_events_checklist.asp
- See also: The PTSD checklist for DSM-5 (PCL-5) — https://www.ptsd.va.gov/professional/assessment/adult-sr/ptsd-checklist.asp